CLINICAL TRIAL: NCT00469638
Title: Ablation Success With the Use of Steerable AGILIS NxT Introducer Compared With Conventionally Used Swartz SL0.
Brief Title: Efficacy and Safety Study on Agilis NxT Introducer in AF Patients
Acronym: AGILIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Alexander Huemmer, St Jude Medical Germany, GMBH
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A07
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; paroxysmal; persistent; symptomatic; ablation; catheter; introducer; Agilis NxT; sinus rhythm; paroxysmal atrial fibrillation; persistent atrial fibrillation; symptomatic atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Agilis sheeth group (Experimental)
  Interventions: Procedure: Left atrial catheter ablation guided by introducer using Agilis sheeth
- Non-steerable sheeth group (Active Comparator)
  Interventions: Procedure: Left atrial catheter ablation guided by introducer using Non-steerable sheeth

INTERVENTIONS:
Procedure: Left atrial catheter ablation guided by introducer using Agilis sheeth — Left atrial catheter ablation guided by introducer using Agilis sheeth
  Arms: Agilis sheeth group
Procedure: Left atrial catheter ablation guided by introducer using Non-steerable sheeth — Left atrial catheter ablation guided by introducer using Non-steerable sheeth
  Arms: Non-steerable sheeth group

SUMMARY:
To prove if the success rate of curative treatment of atrial fibrillation in left atrial circumferential pulmonary vein ablation is higher by using a steerable transseptal introducer giving access to the left atrium then by using a conventionally introducer with fixed curve.

DETAILED DESCRIPTION:
To prove if the success rate of curative treatment of atrial fibrillation in left atrial circumferential pulmonary vein ablation is higher by using a steerable transseptal introducer giving access to the left atrium then by using a conventionally introducer with fixed curve; in patients with paroxysmal or persistent symptomatic Atrial Fibrillation.

Primary Endpoint: rate of patients in stable sinus rhythm at 6 Month Follow Up

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal or persistent symptomatic atrial fibrillation
* Resistant to at least 1 anti arrhythmic drug
* Left atrial diameter less then 60 mm (TTE, parasternal)
* Atrial fibrillation documented by ECG
* Patient is willing and available to perform all Follow Ups

Exclusion Criteria:

* Permanent atrial fibrillation
* Pre existing left atrial fibrillation ablation
* Atrial fibrillation due to reversible cause
* Known intracardiac or other thrombi
* Pregnancy
* Women of child bearing potential without negative pregnancy test within 48 hours prior to ablation
* Contraindication for anticoagulation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
rate of patients in stable sinus rhythm (free of Atrial Fibrillation and Left Atrial Flutter) | 6 months post ablation

SECONDARY OUTCOMES:
rate of patients in stable sinus rhythm (free of Atrial Fibrillation and Left Atrial Flutter) at 3 months post ablation rate of pulmonary vein isolation completely isolated rate of complications procedure duration X-ray duration | 6 month post ablation

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, Prof. Dr., Principal Investigator — Herzzentrum Leipzig, Abteilung für Rhythmologie, Strümpellstraße 39, 04289 Leipzig, Germany
Locations (1):
- Herzzenturm Leipzig, Leipzig, Germany

REFERENCES:
- [Background] Kannel WB, Abbott RD, Savage DD, McNamara PM. Epidemiologic features of chronic atrial fibrillation: the Framingham study. N Engl J Med. 1982 Apr 29;306(17):1018-22. doi: 10.1056/NEJM198204293061703. PMID 7062992
- [Background] Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation as an independent risk factor for stroke: the Framingham Study. Stroke. 1991 Aug;22(8):983-8. doi: 10.1161/01.str.22.8.983. PMID 1866765
- [Background] Piorkowski C, Hindricks G, Weiss S et al: Long term outcome of circumferential left atrial PV ablation using a steerable transseptal sheath. Poster European Society of Cardiology 2006, Barcelona
- [Derived] Piorkowski C, Eitel C, Rolf S, Bode K, Sommer P, Gaspar T, Kircher S, Wetzel U, Parwani AS, Boldt LH, Mende M, Bollmann A, Husser D, Dagres N, Esato M, Arya A, Haverkamp W, Hindricks G. Steerable versus nonsteerable sheath technology in atrial fibrillation ablation: a prospective, randomized study. Circ Arrhythm Electrophysiol. 2011 Apr;4(2):157-65. doi: 10.1161/CIRCEP.110.957761. Epub 2011 Jan 19. PMID 21248246